CLINICAL TRIAL: NCT02852863
Title: Ultrasound Assessment of Changes in Gastric Volume and Content Before and After Chewing Gum
Brief Title: Identification of Changes in Gastric Volume and Content by Ultrasound Before and After Chewing Gum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Jose Alejandro Valencia, MD, Fundación Santa Fe de Bogota
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCEI-5523-2016
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Gastric Volume
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrasound (case only) (Experimental): Subjects will fast for a minimum of 8 hours. Ultrasound assessment of gastric volume and content will determine basal conditions. Next, subjects will chew gum for one hour with changes of gum every 20 minutes (a total of 3 gums will be chewed per subject). Once the last gum is chewed, the gum will be disposed in the trashcan. Three more ultrasound assessments will take place: immediately after one hour of chewing gum, and at the first and second hour after chewing gum has stopped. The content will be classified as empty, with fluids, or with solid. In case of fluids, volume will be measured.
  Interventions: Other: Gum

INTERVENTIONS:
Other: Gum — Subjects will fast for a minimum of 8 hours. A baseline ultrasound assesment will be performed to evaluate gastric content. Next, subjects will chew sugarless gum for one hour with changes of gum every 20 minutes (a total of 3 gums will be chewed per subject). Once the last gum is chewed, the gum will be disposed in the trashcan. Three more ultrasound assessments will take place: immediately after one hour of chewing gum, and at the first and second hour after chewing gum has stopped. The content will be classified as empty, with fluids, or with solid. In case of fluids, volume will be measured.

SUMMARY:
To identify by ultrasound the possible changes in gastric volume and content after chewing gum for an hour in volunteers with complete fasting (more than 8 hours).

ELIGIBILITY:
Inclusion Criteria:

* adults older or equal than 18 years old
* Minimum of 8 hours of fasting
* must work/study at Fundacion Santa Fe

Exclusion Criteria:

* Comorbidities such as obesity, renal failure, diabetes
* Gastrointestinal Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Gastric volume change in mL | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Fundacion SantaFe de Bogota, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Yes